CLINICAL TRIAL: NCT06846892
Title: Comparison of the Effectiveness of Reformer Pilates and Conventional Physiotherapy Rehabilitation Practices in Patients With Lumbar Disc Herniation
Brief Title: Comparison of the Effectiveness of Reformer Pilates and Conventional Physiotherapy in Lumbar Disc Herniation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasemin Şahbaz (Other)
Collaborators: Amasya University (Other); Okan University (Other)
Responsible Party: Sponsor-Investigator, Yasemin Şahbaz, assistant professor, University of Beykent
Organization: University of Beykent (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UBEYKENT-13
Record Dates: First submitted 2025-02-20; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Disc Herniation
Keywords: Reformer Pilates; Conventional Physiotherapy; Lumbar Disc Herniation; Pain Management; Fatigue
MeSH Terms: conditions — Intervertebral Disc Displacement; Agnosia; Fatigue | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Factorial Assignment randomized controlled trial 2 groups
Masking Description: Individuals between the ages of 21-50, who had complaints of low back pain for at least three months and were diagnosed with lumbar disc herniation were included in the study. Inclusion criteria included not having had any spinal surgery in the last six months, regularly attending the program to be implemented, and being able to communicate. Systemic diseases affecting pain such as fibromyalgia, neurological or orthopedic disorders, having received physical therapy in the last eight weeks, the presence of spinal stenosis, spondylolysis, spondylolisthesis or other lumbar degenerative diseases, and pregnancy were determined as exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer Pilates Group (Experimental): The study group participated in a 12-session Reformer Pilates exercise program, performed twice a week, with each session lasting 45-50 minutes. The treatment duration for this group was set to 6 weeks, and the effects of the program on pain management, functional recovery, fatigue, and kinesiophobia were evaluated.
  Interventions: Procedure: Exercise
- Conventional Physiotherapy Group (Active Comparator): The control group, on the other hand, underwent a conventional physiotherapy protocol, with a total of 30 sessions, performed five days a week, and each session lasting 45-50 minutes. This protocol likely included manual therapy, electrotherapy, and exercises. The effects of conventional physiotherapy on pain, fatigue, anxiety, and kinesiophobia were examined. Both groups were assessed before and after treatment using the McGill-Melzack Pain Questionnaire, Fatigue Severity Scale, Pittsburgh Sleep Quality Index, Beck Anxiety Inventory, Tampa Scale of Kinesiophobia, and the SF-36 Quality of Life Scale.
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Exercise — Both groups were given a total of 12 sessions of Williams exercises, two days a week, in 20-minute sessions, accompanied by a physiotherapist. Williams back exercises are an exercise method that aims to increase lumbar flexion and strengthen the abdominal and gluteal muscles. The exercise program included pelvic tilts, single and double knee pulls, partial crunches, hamstring stretches, hip flexor stretches and squats. In addition, the patients continued their Williams exercises at home three days a week.

SUMMARY:
This study aims to examine the effects of Reformer Pilates on patient-reported outcomes such as pain level, fatigue, sleep quality, anxiety, kinesiophobia, and quality of life in individuals with lumbar disc herniation (LDH) and to compare its effectiveness with conventional physiotherapy protocols.

DETAILED DESCRIPTION:
All participants underwent a rehabilitation program for six weeks. Pre- and post-treatment assessments were conducted, and the results of the groups were compared. The Reformer Pilates group participated in a 12-session Pilates exercise program, performed twice a week for 45-50 minutes per session, while the Conventional Physiotherapy group underwent a 30-session conventional physiotherapy program, performed five days a week for 45-50 minutes per session.

Assessment tools included the McGill-Melzack Pain Questionnaire, Fatigue Severity Scale, Pittsburgh Sleep Quality Index, Beck Anxiety Inventory, Tampa Scale of Kinesiophobia, and SF-36 Quality of Life Scale. Measurements were taken twice: before and after treatment.

In post-treatment group comparisons, a significant difference was found in pain levels in the Reformer Pilates group and fatigue levels in the Conventional Physiotherapy group. Within-group analyses showed significant improvements in pain, fatigue, kinesiophobia, and physical function subdomains in the Reformer Pilates group, while the Conventional Physiotherapy group showed significant improvements in fatigue, anxiety, and kinesiophobia scores.

In conclusion, Reformer Pilates was found to be an effective method for pain management, whereas Conventional Physiotherapy provided more notable benefits for fatigue management. Both methods were effective in managing kinesiophobia and fatigue, highlighting the importance of tailoring treatment plans to meet the individual needs of patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 21 and 50 years
* Complaints of low back pain for at least three months
* Diagnosed with lumbar disc herniation
* No spinal surgery in the last six months
* Regular participation in the program
* Ability to communicate
* Exclusion Criteria:
* Presence of systemic diseases affecting pain, such as fibromyalgia
* Presence of neurological or orthopedic disorders
* Receiving physical therapy in the past eight weeks
* Presence of spinal stenosis, spondylolysis, spondylolisthesis, or other lumbar -degenerative diseases
* Pregnancy status

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2024-11-29 (Actual)

PRIMARY OUTCOMES:
McGill Pain Questionnaire | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The McGill Pain Questionnaire is a reliable tool used to assess pain in a multifaceted way. It addresses the sensory (11 words), emotional (5 words), and general intensity dimensions of pain. Patients select appropriate words that describe their pain to create a total pain score. Pain intensity is measured using a 6-point Likert scale (0 = no pain, 5 = unbearable) and a 10 cm Visual Analog Scale (VAS). This questionnaire is an effective method for evaluating both the intensity and qualitative dimensions of pain.
Tampa Scale of Kinesiophobia | Baseline (pre-treatment) and 6 weeks (post-treatment)
  This scale is a 17-item tool that evaluates activity-related injury, injury recurrence, fear, and avoidance. It is used in musculoskeletal disorders (such as low back pain, fibromyalgia). Scores range from 17 to 68, with higher scores indicating a higher level of kinesiophobia.
SF-36 Quality of Life Scale | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The SF-36 is an internationally standardized questionnaire used to assess health status and satisfaction, with a structure suitable for different patient groups. The questionnaire analyzes an individual's functional status under eight main categories: social functioning, cognitive health, physical functioning, pain, emotional resilience, energy/vitality, general health perception, and physical health. Each subscale has a different scoring system, and higher scores indicate better health and improved quality of life.
Beck Anxiety Inventory | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The BAI is a 21-item Likert-type scale developed by Beck in 1961 to assess depressive symptoms. Each item is scored between 0 and 3, and the total score ranges from 0 to 63. Higher scores indicate more severe levels of depression.
Pittsburgh Sleep Quality Index | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The PSQI is a 19-item scale used to assess sleep quality over the past month. It was developed by Buysse and colleagues in 1989. The scale is divided into 7 subcomponents, each scored between 0 and 3. The total score ranges from 0 to 21, with scores above 5 indicating poor sleep quality.
Fatigue Severity Scale | Baseline (pre-treatment) and 6 weeks (post-treatment)
  The FSS is a 9-item scale used to assess fatigue. Items are rated on a scale from 1 to 7, and the total score is divided by 9 to calculate the average score. An average score of <4 indicates no fatigue, while a score of ≥4 indicates the presence of fatigue.

CONTACTS AND LOCATIONS:
Locations (1):
- Yasemin Şahbaz, Beyli̇kdüzü, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yakut Y, Yakut E, Bayar K, Uygur F. Reliability and validity of the Turkish version short-form McGill pain questionnaire in patients with rheumatoid arthritis. Clin Rheumatol. 2007 Jul;26(7):1083-7. doi: 10.1007/s10067-006-0452-6. Epub 2006 Nov 15. PMID 17106618
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Buysse DJ, Hall ML, Strollo PJ, Kamarck TW, Owens J, Lee L, Reis SE, Matthews KA. Relationships between the Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), and clinical/polysomnographic measures in a community sample. J Clin Sleep Med. 2008 Dec 15;4(6):563-71. PMID 19110886
- [Background] Armutlu K, Korkmaz NC, Keser I, Sumbuloglu V, Akbiyik DI, Guney Z, Karabudak R. The validity and reliability of the Fatigue Severity Scale in Turkish multiple sclerosis patients. Int J Rehabil Res. 2007 Mar;30(1):81-5. doi: 10.1097/MRR.0b013e3280146ec4. PMID 17293726